CLINICAL TRIAL: NCT06386380
Title: Adversity and Its Association With the Development and Expression of Rheumatic Diseases
Acronym: RD
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Dr, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE-4906
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: RhA - Rheumatoid Arthritis
Keywords: Adversity; Rheumatic diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases | interventions — ametantrone; Cyclin-Dependent Kinase Inhibitor p16; Cellular Senescence

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A 10 ml peripheral blood sample will be taken by venipuncture with the Vacutainer® system in tubes with EDTA anticoagulant. DNA will be extracted using the commercial Wizard® system (Promega TM cat: A1620) based on salt precipitation. The extracted DNA will be quantified in a Nanodrop spectrophotometer, diluted, and preserved at -20°C until use. The Institute's Cellular Immunology and Genetics laboratories will analyze the DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rheumatoid arthritis: Patients with rheumatoid arthritis outpatients from the National Institute of Medical Sciences
  Interventions: Other: Rheumatic diseases Mistreatment Scale (RDMS); Other: Routine assessment of patient index data 3 (RAPID-3); Other: Health Assessment Questionnaire (HAQ); Other: WHOQOL-BREF; Other: Depression, Anxiety and Stress Scale (DASS-21); Other: Brief Resilient Coping Scale; Genetic: Expression of CDKN2A /p16INK4a; Other: Immunophenotype of leukocyte subpopulations; Genetic: Telomere length; Other: Cellular senescence

INTERVENTIONS:
Other: Rheumatic diseases Mistreatment Scale (RDMS) — In 2012, Giraldo-Rodríguez developed and validated the Geriatric Mistreatment Scale (GAS); translation, cultural adaptation, and validation were performed prior to its application.
  Other Names: RD-MS
Other: Routine assessment of patient index data 3 (RAPID-3) — RAPID- 3 measures: function, pain, and patient global status estimate. Each of the three individual measures is scored 0 to 10, for a total of 30
  Other Names: RAPID-3
Other: Health Assessment Questionnaire (HAQ) — The HAQ is based on five patient-centered dimensions: disability, pain, medication effects, costs of care, and mortality.
  Other Names: HAQ
Other: WHOQOL-BREF — WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health, psychological health, social relationships, and environmental health; it also contains QOL and general health items
Other: Depression, Anxiety and Stress Scale (DASS-21) — DASS-21 is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains seven items, divided into subscales with similar content.
  Other Names: DASS-21
Other: Brief Resilient Coping Scale — The Brief Resilient Coping Scale is a 4-item measure designed to capture tendencies to cope with stress in a highly adaptive manner.
  Other Names: BRCS
Genetic: Expression of CDKN2A /p16INK4a — CDKN2A/p16INK4a expression will be measured using the Taqman qPCR assay (TaqMan Universal Master Mix II, with UNG, Applied Biosystems, Foster City, USA) according to the manufacturer's specifications.
Other: Immunophenotype of leukocyte subpopulations — CD4+ and CD8+ subpopulations will be analyzed. Blood samples will be analyzed by 8-color flow cytometry (Becton Dickinson Canto II cytometer) using fluorescently labeled antibodies from Biolegend Inc. (San Diego, USA).
Genetic: Telomere length — The rLTL will be estimated by quantitative monochromatic multiplex PCR (MM-qPCR). Integrated DNA Technologies, Inc. (IDT, Coralville, IA, USA) will synthesize the primers used for telomere measurements.
Other: Cellular senescence — Expression of co-stimulatory molecules and surface receptors CD27- and CD28-

SUMMARY:
Epidemiological evidence shows that adverse experiences, particularly, but not exclusively in childhood, are predictors of poor long-term health outcomes and certain social domains. In the field of rheumatic diseases, traumatic events, not only in childhood, have been associated with hospitalization, chronic pain, inflammation, worse outcomes, severity of the disease, and mortality. Some mechanisms proposed to explain the association between the experience of adversity and the development of chronic diseases include an impact on the physiology of immune system cells, gene expression due to DNA modification, and cellular senescence.

With this background, the investigators wonder if, for patients with rheumatoid arthritis, the presence of adversity understood as a history of violence in childhood and abuse due to suffering from rheumatoid arthritis is associated with markers of cellular senescence and with the severity of illness.

DETAILED DESCRIPTION:
To answer this question, the investigators proposed conducting a study on outpatients diagnosed with rheumatoid arthritis treated at the INCMNSZ.

Patients who agree to participate will be asked to answer some questionnaires to report their perception of child abuse and abuse derived from suffering from rheumatoid arthritis, disease activity, disability, quality of life, anxiety, stress, depression, and resilience.

Additionally, a peripheral blood sample will be taken to evaluate cellular senescence through CD27, CD28, and CD57 expression, the relative expression of the p16INK4a gene in CD3+ lymphocytes, HLA-DR, CD25, and CD69, and telomere length. Finally, the expression of the severity of the disease will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a rheumatoid arthritis diagnosis, according to their primary rheumatologist who agrees to participate

Exclusion Criteria:

* Patients with a not confirmed rheumatoid arthritis diagnosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with rheumatoid arthritis outpatients from the National Institute of Medical Sciences
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Adversity and senescence in patients with rheumatoid arthritis | At inclusion (baseline moment) (cross-sectional study)]
  To evaluate whether the presence of adversity (history of abuse in childhood and/or abuse associated with RD) is associated with markers of senescence in patients with rheumatoid arthritis.

SECONDARY OUTCOMES:
Eexpression of the p16INK4a gene in CD3+ | At inclusion (baseline moment) (cross-sectional study)]
  Compare the relative expression of the p16INK4a gene in CD3+ lymphocytes between rheumatoid arthritis patients with and without adversity.
Telomere length | At inclusion (baseline moment) (cross-sectional study)]
  Compare telomere length between RA patients with and without adversity.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia MD Pascual-Ramos, MD, Principal Investigator — IInstituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baumer Y, Powell-Wiley TM. Interdisciplinary approaches are fundamental to decode the biology of adversity. Cell. 2021 May 27;184(11):2797-2801. doi: 10.1016/j.cell.2021.04.010. PMID 34048701